CLINICAL TRIAL: NCT05382390
Title: Dual Growth Factor (rhTPO + G-CSF) and Chemotherapy Combination Regimen in Acute Myeloid Leukemia: Study Protocol for a Randomized Controlled Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huihan Wang (Other)
Responsible Party: Sponsor-Investigator, Huihan Wang, Deputy Chief Physician, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hhhWang
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Aclarubicin; Granulocyte Colony-Stimulating Factor; Cytarabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To compensate for the need for an open-label design, the primary outcome data are collected with blinding. The staff responsible for data monitoring and statistician will also be blinded to the treatment groups until the statistical analysis was finalized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lderly Patients With Acute Myeloid Leukemia DCTAG (Experimental): decitabine (15 mg/m2 daily, days 1-5); low-dose cytarabine (10 mg/m2 q12 h, days 3-9); rhTPO (15,000 U daily, days 2, 4, 6, 8, and 10-24 or until a platelet count > 50 × 109/L was observed); aclarubicin (14 mg/m2 daily, days 3-6); and G-CSF (300 μg daily, days 2-9).
  Interventions: Drug: rhTPO; Drug: Decitabine
- lderly Patients With Acute Myeloid Leukemia (Other): decitabine (15 mg/m2 daily, days 1-5); low-dose cytarabine (10 mg/m2 q12 h, days 3-9); aclarubicin (14 mg/m2 daily, days 3-6); and G-CSF (300 μg daily, days 2-9).
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: rhTPO — decitabine (15 mg/m2 daily, days 1-5); low-dose cytarabine (10 mg/m2 q12 h, days 3-9); rhTPO (15,000 U daily, days 2, 4, 6, 8, and 10-24 or until a platelet count > 50 × 109/L was observed); aclarubicin (14 mg/m2 daily, days 3-6); and G-CSF (300 μg daily, days 2-9).
  Other Names: Decitabine; Aclarubicin; G-CSF; Cytarabine
  Arms: lderly Patients With Acute Myeloid Leukemia DCTAG
Drug: Decitabine — decitabine (15 mg/m2 daily, days 1-5); low-dose cytarabine (10 mg/m2 q12 h, days 3-9); aclarubicin (14 mg/m2 daily, days 3-6); and G-CSF (300 μg daily, days 2-9).
  Other Names: Aclarubicin; G-CSF; Cytarabine

SUMMARY:
Acute myeloid leukemia (AML) is a disease affecting older adults, although optimal strategies for treating such patients remain unclear. This prospective phase II, openlabel, multicenter study was designed to assess the efficacy and safety of two hematologic growth factors, recombinant human thrombopoietin (rhTPO) and granulocyte colonystimulating factor (G-CSF), in combination with decitabine, cytarabine, and aclarubicin (D-CTAG regimen) to treat older adults with newly diagnosed AML (Identifier: NCT04168138). The above agents were administered as follows: decitabine (15 mg/m2 daily, days 1-5); low-dose cytarabine (10 mg/m2 q12 h, days 3-9); rhTPO (15,000U daily, days 2, 4, 6, 8, 10-24 or until >50×109/L platelets); aclarubicin (14 mg/m2 daily, days 3-6); and G-CSF (300 μg daily, days 2-9). We concurrently monitored historic controls treated with decitabine followed by cytarabine, aclarubicin, and G-CSF (D-CAG) only. After the first D-CTAG cycle, the overall response rate (ORR) was 84.2% (16/19), including 13 (73.7%) complete remissions (CRs) and three (15.8%) partial remissions. This CR rate surpassed that of the D-CAG treatment (p < 0.05). Median overall survival (OS) time in the D-CTAG group was 20.2 months (range, 4-31 months), compared with 14 months in the D-CAG group, and 1-year OS was 78%. The proportion of those experiencing grade III-IV thrombocytopenia was significantly lower for D-CTAG (57.9%) than for D-CAG (88.4%; p < 0.05). Ultimately, the curative effect of adding rhTPO was not inferior to that of D-CAG, and D-CTAG proved safer for elderly patients, especially in terms of hematologic toxicity. A prospective phase III randomized study is warranted to confirm these observations.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is one of the most common hematologic malignancies and affects older adults. The median age at diagnosis is 67 years. As the elderly increasingly account for a greater population percentage, AML is becoming more problematic. During the past 30 years, outcomes have improved for younger patients, whereas the prospects for older adults (> 60 years) have remained poor. The response rate in older adults given standard induction regimens is < 50%, and median overall survival (OS) is < 1 year. Older adults elderly are also inordinately burdened by unfavorable cytogenetic defects, medical comorbidities, and reduced tolerability to intensive chemotherapeutic protocols. These vulnerabilities predispose older adults to poorer outcomes than their younger counterparts, conferring lower response rates and shortened survival times (progression-free and overall survival [OS]). Safe and effective treatments for elderly patients with AML are thus urgently needed.

In 2000, Saito et al introduced a regimen of granulocyte colony-stimulating factor (G-CSF) plus low-dose cytarabine (ara-C) and aclarubicin (ACR) for use in this setting (CAG regimen), in an attempt to incorporate a hematologic growth factor in AML induction therapy, rather than relying on supportive care. The addition of decitabine, a demethylation agent, further improved the prognosis, yielding a 10-month median OS. This successful use of G-CSF in an induction regimen for AML confirmed its utility, helping to increase efficacy and reduce side effects in elderly patients.

Thrombopoietin (TPO) is a major factor in regulating megakaryocytic proliferation, maturation, and platelet formation. Recombinant human TPO (rhTPO) has been approved by China's State Food and Drug Administration to treat thrombocytopenia after chemotherapy. TPO and c-MPL receptors are also involved in various physiologic processes, such as mitigating myocardial injury, nerve repair, vascular regeneration, sex hormone secretion, and immune regulation. However, the role of rhTPO in an induction regimen for AML is unreported as yet.

To determine if adding rhTPO to D-CAG (G-CSF) will increase the overall response rate (ORR) while decreasing the side effect of toxic agents, we designed a regimen of rhTPO and G-CSF in combination with decitabine, cytarabine, and aclarubicin (D-CTAG regimen). This trial aimed to determine the safety and efficacy of this D-CTAG regimen as a treatment for older adult patients with newly diagnosed AML.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or above, male or female; Acute Myeloid Leukemia (non-M3) diagnosed according to the 2008 World Health Organization (WHO) diagnostic criteria for myeloid malignancies; Newly diagnosed, no treatment for anti-leukemia; The Eastern Cooperative Oncology Group（ECOG） status score is 0 to 3 points; Expected survival time ≥ 3 months; No serious heart, lung, liver or kidney disease; History of no thromboembolism Ability to understand and be willing to sign the informed consent form of this trial.

Exclusion Criteria:

* used to be allergic to the drugs contained in the protocol or to drugs similar in chemical structure to the test drugs; serious active infections; Patients with extramedullary lesions; Patients who use drugs and long-term alcohol abuse to influence the evaluation of test results; Inability to obtain informed consent and cannot complete the trial treatment and examination procedures because of mental illness or other conditions Patients with clinically significant corrected QT interval (QTc) prolongation (male > 450ms, female > 470ms), Ventricular Tachycardia (VT), Atrial Fibrillation (AF), grade II or higher heart block, Myocardial Infarction (MI) within 1 year, Congestive Heart Failure (CHF), coronary heart disease with symptoms who need medical treatment; Abnormal liver function (total bilirubin > 1.5 times the upper limit of normal value, Alanine aminotransferase(ALT) / Aspartate aminotransferase (AST) >2.5 times the upper limit of normal value or ALT / AST in patients with liver invasion > 5 times the upper limit of normal value of normal), abnormal renal function (serum Creatinine > 1.5 times the upper limit of normal); The investigator determine that the participants are not suitable

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-01-21 (Estimated); Study Completion 2026-01-21 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 2 years after the end of treatment of the last patient enrolled
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- ShengJing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No